CLINICAL TRIAL: NCT03671031
Title: Isolated Roux Loop Versus Conventional Pancreaticojejunostomy Following Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Egemen Ozdemir, Principal Investigator, Inonu University
Other Study IDs: 2018/16-22
Record Dates: First submitted 2018-09-11; First posted 2018-09-14 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Pancreatic Fistula
Keywords: pancreatic fistula; pancreatic leak; whipple operation; roux-en-y
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- isolated roux loop: isolated roux loop reconstruction following pancreaticoduodenectomy as the first group.
  Interventions: Procedure: isolated roux loop
- single loop: single loop reconstruction following pancreaticoduodenectomy as the second group.
  Interventions: Procedure: single loop

INTERVENTIONS:
Procedure: isolated roux loop — Isolated roux loop reconstruction following pancreaticoduodenectomy
  Groups: isolated roux loop
Procedure: single loop — Conventional single loop reconstruction following pancreaticoduodenectomy
  Groups: single loop

SUMMARY:
Pancreaticoduodenectomy is a commonly applied operation for the treatment of benign and malignant diseases of periampullary region. Although recent progress in surgical techniques and medical care reduced the mortality rate of this operation below 5% in some institutes, the morbidity rate still remains high as 40-50% (1,2). Pancreatic anastomotic leaks and fistulas continue to be the main source of morbidity and mortality after pancreaticoduodenectomy. Although there are several recommended techniques to reduce the rate of pancreatic fistulas, optimal pancreatic reconstruction technique is still controversial (3-5). One of the recommended techniques for pancreatic reconstruction is isolated Roux loop pancreaticojejunostomy (6). With this method, as pancreatic anastomosis is kept away from biliary and gastric anastomoses, activation of the pancreatic enzyme precursors is blocked and in this way a reduction in the rate and severity of pancreatic fistula and also in the overall morbidity and mortality can be achieved (6-8).

In this study, it is aimed to examine if isolated Roux loop pancreaticojejunostomy is superior to conventional pancreaticojejunostomy on postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent pancreaticoduodenectomy.

Exclusion Criteria:

* patients with missing data
* patients who underwent total pancreatectomy
* patients who had pancreaticogastrostomy as the reconstruction method
* patients who had emergency pancreaticoduodenectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who underwent pancreaticoduodenectomy at General Surgery Clinic in Inonu University between January 2009 and June 2018
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Severity of postoperative pancreatic fistula | 1 week
  Assessed according to International Study Group on Pancreatic Fistula definition

SECONDARY OUTCOMES:
Rate of postoperative pancreatic fistula | 1 week
  Number of participants with postoperative pancreatic fistula
Operation time | 1 week
  in minutes
Duration of hospital stay | 1 week
  in days
Duration of intensive care unit stay | 1 week
  in days
30-day mortality | 1 week
  Number of participants died in 30 days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Egemen Ozdemir, MD, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang YM, Tian XD, Zhuang Y, Wang WM, Wan YL, Huang YT. Risk factors of pancreatic leakage after pancreaticoduodenectomy. World J Gastroenterol. 2005 Apr 28;11(16):2456-61. doi: 10.3748/wjg.v11.i16.2456. PMID 15832417
- [Background] El Nakeeb A, Salah T, Sultan A, El Hemaly M, Askr W, Ezzat H, Hamdy E, Atef E, El Hanafy E, El-Geidie A, Abdel Wahab M, Abdallah T. Pancreatic anastomotic leakage after pancreaticoduodenectomy. Risk factors, clinical predictors, and management (single center experience). World J Surg. 2013 Jun;37(6):1405-18. doi: 10.1007/s00268-013-1998-5. PMID 23494109
- [Background] Reid-Lombardo KM, Farnell MB, Crippa S, Barnett M, Maupin G, Bassi C, Traverso LW; Pancreatic Anastomotic Leak Study Group. Pancreatic anastomotic leakage after pancreaticoduodenectomy in 1,507 patients: a report from the Pancreatic Anastomotic Leak Study Group. J Gastrointest Surg. 2007 Nov;11(11):1451-8; discussion 1459. doi: 10.1007/s11605-007-0270-4. Epub 2007 Aug 21. PMID 17710506
- [Background] Wente MN, Shrikhande SV, Muller MW, Diener MK, Seiler CM, Friess H, Buchler MW. Pancreaticojejunostomy versus pancreaticogastrostomy: systematic review and meta-analysis. Am J Surg. 2007 Feb;193(2):171-83. doi: 10.1016/j.amjsurg.2006.10.010. PMID 17236843
- [Background] Xiong JJ, Altaf K, Mukherjee R, Huang W, Hu WM, Li A, Ke NW, Liu XB. Systematic review and meta-analysis of outcomes after intraoperative pancreatic duct stent placement during pancreaticoduodenectomy. Br J Surg. 2012 Aug;99(8):1050-61. doi: 10.1002/bjs.8788. Epub 2012 May 24. PMID 22622664
- [Background] Machado MC, da Cunha JE, Bacchella T, Bove P. A modified technique for the reconstruction of the alimentary tract after pancreatoduodenectomy. Surg Gynecol Obstet. 1976 Aug;143(2):271-2. PMID 941087
- [Background] Kingsnorth AN. Safety and function of isolated Roux loop pancreaticojejunostomy after Whipple's pancreaticoduodenectomy. Ann R Coll Surg Engl. 1994 May;76(3):175-9. PMID 7912489
- [Background] Albertson DA. Pancreaticoduodenectomy with reconstruction by Roux-en-Y pancreaticojejunostomy: no operative mortality in a series of 25 cases. South Med J. 1994 Feb;87(2):197-201. doi: 10.1097/00007611-199402000-00010. PMID 8115883